CLINICAL TRIAL: NCT00957606
Title: Osteoporosis Among Men Treated With Androgen Deprivation for Prostate Cancer: Symptoms, Risc Factors, and Prevention
Brief Title: Osteoporosis Among Men Treated With Androgen Deprivation for Prostate Cancer
Acronym: Osteoporosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Mads Hvid Poulsen, MD, Department of Urology, Odense University Hospital, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCa & Osteoporosis 09; S-20080004
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Prostate Cancer; Androgen Deprivation Therapy; Osteoporosis
Keywords: Prostate cancer; androgen deprivation therapy; osteoporosis
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis | interventions — Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: blood sampling, DXA-scan, bone scintigraphy — Blood sampling 5 times DXA-scan 5 times Bone scintigraphy 3 times

SUMMARY:
The purpose of this study is

* to determine the rate of osteoporosis among patients with advanced prostate cancer.
* to propose an algorithm for early detection of patients with advanced prostate cancer who are at risk of developing osteoporosis.

DETAILED DESCRIPTION:
Patients with advanced prostate cancer are included at the initiating of androgen deprivation therapy.

The patients are followed for 2 years after inclusion with blood sampling, DXA-scan, questionnaire, bone scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer
* Initiation of androgen deprivation therapy
* Oral and written informed consent

Exclusion Criteria:

* They withdraw their consent
* Treatment for osteoporosis within the last year
* Other malignancy
* Other bone disease, bedbound, use of steroid

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis, either T-score < -2,5 or osteoporosis fracture | 2½ years

CONTACTS AND LOCATIONS:
Overall Officials: Mads H Poulsen, MD, Principal Investigator — Department of Urology, Odense University Hospital, Denmark; Steen Walter, MD, DMSci, Professor, Study Chair — Department of Urology, Odense University Hospital, Denmark; Morten MF Nielsen, MD, Study Chair — Department of Endocrinology, Odense University Hospital, Denmark; Kim Brixen, MD, PhD, Professor, Study Chair — Department of Endocrinology, Odense University Hospital, Denmark; Claus Dahl, MD, Study Chair — Department of Urology, Roskilde Hospital, Denmark; Peter Eskildsen, MD, DMSci, Study Chair — Department of Endocrinology, Køge Hospital, Denmark; Oke Gerke, PhD, Study Chair — University of Southern Denmark; Bo Abrahamsen, MD, PhD, Professor, Study Chair — Faculty of Health Sciences, University of Southern Denmark, Denmark
Locations (2):
- Denmark (2):
  - Department of Urology, Odense University Hospital, Odense
  - Department of Urology, Roskilde Hospital, Roskilde